CLINICAL TRIAL: NCT04722497
Title: HSR200262-Effectiveness of a Visual Noise Warning System on Noise Levels in the Labor and Delivery Operating Room: A Quality Improvement Program
Brief Title: Noise in the OR: A Quality Improvement Program
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Megan Whitham, MD, Maternal Fetal Medicine fellow, University of Virginia
Other Study IDs: HSR200262
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Noise; Adverse Effect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physicians and nurses: All physicians, nurses, involved in a cesarean births are included in the cohort.
  Interventions: Other: Sound Education
- Patients undergoing cesarean births: All patients undergoing cesarean births

INTERVENTIONS:
Other: Sound Education — All physicians and nurses involved in cesarean births will be given an education intervention explaining the impact of noise levels on stress and focus. The SoundEar device will be used as an intervention tool to inform operating room physicians and nurses when the noise level is above the desired level.
  Groups: Physicians and nurses

SUMMARY:
During Phase I, disguised SoundEar noise devices will be used to record the noise levels in the operating rooms on Labor and Delivery during Cesarean births. Survey data will be acquired from physicians, nurses, and patients to determine if the sound in the operating rooms during surgery impacted the stress levels of those involved. An educational intervention will then be held for the physicians and nurses, and Phase II will involve having the SoundEar devices exposed. When the sound level reaches a distracting level, the light on the device will change to bright red. Surveys will be collected to determine if there is a difference in the stress levels if and when the noise level in the operating room is decreased during cesarean births.

DETAILED DESCRIPTION:
For noise measurement and visual feedback, a SoundEar III device will be used. The SoundEar is the most studied and supported AV device maker in medical literature, with option of recording and providing visual feedback, designed specifically to "create awareness about noise". The device measures the environmental sound continuously and is also able to provide visual feedback indicating the actual sound level and has been extensively studied for uses in the clinical setting.

The technical specifications of the device are as follows: frequency range 20Hz to 16kHz and scope of measurement of 45dB(A) (similar to bird calls) to 115dB(A) (a sound level that can be encountered at a live rock music venue). The system provides optical feedback in 3 categories: green light (acceptable noise level), orange light (noise level is near the limit) and red light (noise level has exceeded the limit).

The L&D ORs will be equipped with a sound measurement feedback device mounted on the wall visible from the foot end of the operating table. Noise recording can be conducted continuously for 24 hours a day, and downloaded, stored and analyzed weekly. The recorded sound level data can be time-matched with corresponding operations during time stamps.

The study will be divided into 4 phases.

Initially, a baseline validated Weinstein Noise Sensitivity questionnaire (WNS-6B) for subjective noise sensitivity will be collected for all potentially included primary resident surgeons9 as the variability in noise annoyance/disturbance is often best explained by individual subjective noise sensitivity than true noise level.

In phase 1, over a 4-6 month period, we will measure noise decibel level with the noise meter continuously with the optical feedback function concealed and pair this with all scheduled and unscheduled C-sections in the L&D OR. The surgical team members will not specifically be told that data is being collected for a study, but the SoundEar devices will be visible to the surgical team during this phase. We will then plan to collect brief scale questionnaires on a visual analog scale adapted from Engelmann, et al. for all included study cases from the primary resident surgeon, the circulating RN and the patient regarding perceived noise level, stress level and overall experience. . Health care team members will serve as their own nested controls and thus the questionnaires will be de-identified and paired with a unique study ID number generated for each participant---- please note that the first page will only ask for the respondent's name and the questionnaire on the second page will not contain identifying information with the intention of removing the respondents name after their unique identifier has been transcribed to the questionnaire. These cases will serve as nested controls with each provider submitting a response serving as their own baseline control during statistical analysis and will be able to be linked to operative details and patient's chart from date and time noted for the delivery by the respondent. No identifying patient information will be collected on any of the paper questionnaires. Details about: case length, number of attendees in the operating room, blood loss, intraoperative complications, NICU involvement, NICU admission, maternal and neonatal length of stay, postoperative complications, readmissions, and reoperations will be obtained from the patient's chart in a prospective manner.

Each patients who consents to be in the study will complete one questionnaire. The patient will be informed that we are recording the noise levels in the OR during their surgery, and that we are studying the impact of noise levels in the OR on patient and physician stress levels and surgical outcomes.

Examples of the questionnaires are included with this application. The primary RN will also record the case type (scheduled, unplanned, urgent, or emergent), date and case start and stop time for time stamp reference, number of staff members in the L&D OR and pertinent pediatric outcome data (APGAR, gestational age, NICU admission) in his/her portion of the survey. These cases will serve as "controls" and baseline noise data.

A two week washout period will then be planned during which no data will be collected. A difference in noise reduction of 3dB(A) is an important noise level reduction level as it represents a 50% reduction in perceived noise levels. A power calculation can be performed after phase 1 to calculate needed cases to demonstrate a statistical difference in noise reduction with intervention. From the literature, with an average decibel level of roughly 60 dB, and S.D. of 10 dB, 87 cases would be required to demonstrate statistical significance at 80% power.

In phase 2, the visual feedback function will be activated on the noise meters. Providers will be aware of the introduction of the device but receive no formal noise reduction education or knowledge that a study is being conducted in this phase. A threshold of ≤60dB(A) is generally accepted as an "acceptable" level and ≥65dB(A) as an excessive noise level based on the system providers recommendations and per results from previous studies in the medical literature. Optical feedback can then be accordingly activated in these 3 ranges (green light ≤60dB(A), orange light from 60-65dB(A), red light ≥65dB(A)). Similarly, we will collect overall noise data continuously during phase 2 and pair this with all scheduled and unscheduled C-sections in the L&D OR with questionnaire data collected for comparison to the pre-intervention period.

For statistical analysis, surgeons and RN team members will be compared in nested control manner from the preintervention to postintervention time periods with planned sub-analysis of "high-responders" and "low-responders" from results of their previously obtained subjective WNS-6B questionnaires.

After data collection for phase 2, a phase 3 and 4 intervention period may be planned with intervening washout periods. These phases will take place after a 2 week formal education program on noise reduction, combined with the visual feedback function first disabled and then enabled with similar recording of continuous noise decibel level and survey data. The purpose of phase 3 and 4 will be in comparing outcomes from simple introduction of the device versus combined education program on noise awareness. The noise awareness program will also include a prompt that incorporation of noise reduction efforts are ongoing during preoperative time out. Initial sub-analysis of phase 1&2 data should be planned for evaluating efficacy of the visual feedback device alone at improvement in noise outcomes (manuscript #1). Surgical and pediatric outcomes data will also be measured during all time periods for evaluation.

If the intervention is successful at improvement in surgeon stress or patient outcomes, the AV feedback noise meters may be considered for long term adoption into the L&D ORs and future investigation of effectiveness in the Labor and Delivery Room (LDR) during vaginal births could be planned.

ELIGIBILITY:
Inclusion Criteria: the resident surgeon who performs a cesarean section, the resident anesthesiologist, the attending OBGYN and Anesthesiologist, the nurse who is the primary nurse for the patient, and the patient who is undergoing a cesarean section

Exclusion Criteria:At the nurse/physician's discretion, any patient who has suffered a fetal loss or has another serious complication that causes too much stress to expect them to participate in the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the resident surgeon who performs a cesarean section, the resident anesthesiologist, the attending OBGYN and Anesthesiologist, the nurse who is the primary nurse for the patient, and the patient who is undergoing a cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reducing Noise Levels in the Operating Room | 1 year
  Our primary outcome to measure will be noise decibel level over the study time period with a primary end-point of a 3 point reduction in noise decibel level which represents a reduction of 50% perceived noise level.We plan to use univariate and multivariate analysis for our primary outcomes measures of noise reduction.

SECONDARY OUTCOMES:
Noise Disturbance in the Operating Room | 1 year
  Our secondary measured outcomes will be a significant measurable reduction in patient and healthcare team member noise disturbance as measured by Likert scale questionnaires targeting OR experience.We will use ranked match sums for survey analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Megan J Whitham, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No